CLINICAL TRIAL: NCT00914199
Title: Stenting of Coronary Artery Stenoses With Significant Side Branches. Should we, or Should we Not, Perform Dilatation of the Side Branch Through the Main Vessel Stent, if There is Acceptable Blood Flow in the Side Branch?
Brief Title: The Nordic Bifurcation Study III
Acronym: BIF III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evald Hoej Christiansen (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor-Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20070005
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: PCI; Bifurcation lesion
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kissing balloon post-dilatation (Experimental): Percutaneous coronary intervention with implantation of stent using kissing balloon dilatation
  Interventions: Procedure: Percutaneous coronary intervention (PCI)
- No kissing balloon post-dilatation (Experimental): Percutaneous coronary intervention with implantation of stent and not using kissing balloon postdilatation
  Interventions: Procedure: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Implantation of coronary stent in bifurcation lesion.
  Other Names: Percutaneous coronary intervention technique; PCI; PTCA

SUMMARY:
Should we, or should we not, perform dilatation of the side branch through the main vessel stent, if there is acceptable blood flow in the side branch?

DETAILED DESCRIPTION:
Design:

* Randomised open multicentre trial

Patients:

* Number 477

Randomisation:

* Treatment strategy kissing or no kissing balloon post-dilatation

Primary end point:

* Combined end point of: cardiac death, index lesion myocardial infarction, stent thrombosis or target lesion revascularisation after 6 months.

Secondary end points:

* Clinical
* MACE (cardiac death, myocardial infarction, stent thrombosis or target vessel revascularisation) during hospital period, after 1, 8, and 14 months, 2, 3 and, 5 years.
* Cardiac death during hospital period, after 1, 8 and 14 months, 2, 3 and, 5 years.
* Myocardial infarction during hospital period, after 1, 8 and 14 months, 2, 3 and, 5 years.
* Stent thrombosis during hospital period, after 1, 8 and 14 months, 2 and 3 years.
* Target vessel revascularisation during hospital period, after 1, 8 and 14 months, 2 and 3 years.
* Total mortality during hospital period, after 1, 6, 8 and 14 months, 2 and 3 years.
* Target lesion revascularisation during hospital period, after 1, 8 and 14 months, 2 and 3 years.
* Myocardial infarction related to the index procedure.
* CCS angina score after 1, 8 and 14 months, 2, 3 and, 5 years.
* Angiographic. Angiographic significant stenosis (>50%) of main vessel and/or occlusion of the side branch after 8 months.
* Late loss of main vessel and side branch after 8 months.
* Angiographic significant stenosis (>50%) of main vessel and/or side branch after 8 months.
* Angiographic significant stenosis (>50%) of main vessel after 8 months.
* Angiographic significant stenosis (>50%) of side branch after 8 months.
* Markers. All patients with stable angina pectoris and the patients with unstable angina pectoris, who have normal markers (CK-MB or TnT/TnI) before and after the procedure, will enter into the marker study.

End point evaluation:

* Primary and secondary end points will be assessed by an independent end point committee. The end point committee will consist of experienced cardiologists. The detailed end point definitions are the following:
* Q wave myocardial infarction. Appearance of a new Q wave in two or more contiguous leads on ECG.
* Non Q wave myocardial infarction.Infarction, which is considered present in a patient having clinical, angiographic electrocardiographic and/or laboratory evidence of myocardial necrosis with an ECG showing no new Q waves
* Procedure related myocardial infarction. A > threefold increase of CK-MB or Troponin-T/I.
* Target lesion revascularization. Coronary bypass operation with grafting or PCI of index lesion.
* Target vessel revascularization. Coronary bypass operation with grafting or PCI of index vessel
* Stent thrombosis. Stent thromboses are categorized as acute, sub acute, late and very late and as definite, probable and possible (see appendix).
* Vessel measurement. Proximal reference diameter: Vessel diameter proximal to lesion.Distal reference diameter: Vessel diameter distal to lesion.Percentual diameter stenosis: (Reference diameter - minimal luminal diameter)/reference diameter in percent.
* Angiographic restenosis. > 50% diameter stenosis.
* Recommendations for re-revascularization. Main vessel:Angina pectoris, CCS 1 related to index lesion and stenosis diameter >40%* Stenosis diameter >70%*. Side branch: AP, CCS >1 related to index lesion and stenosis diameter >40%*

  * The stenosis diameter is evaluated by eyeballing.

Angiographic core lab:

* The index and follow-up angiograms will be asses by the QCA-laboratories at Department of Cardiology, Paul Stradins Clinical Hospital, Riga, Latvia and Department of Cardiology B, Aarhus University Hospital Skejby, Aarhus N, Denmark.

Definition of index angiography:

* The angiography obtained during the PCI-procedure will be used as index angiography

Follow-up angiography:

* After 8 months conventional diagnostic angiography will be performed and the projections used at the index angiography will be repeated after 0.1 mg intracoronary nitroglycerine. The index angiograms will be stored on CD and sent by mail to the angiographic core laboratories.

Steering committee:

* The steering committee members will be selected on basis of participation in the study. All steering committee members will have full access to the database and will participate in the interpretation of data.

Progress of the study:

* The progress of the study will be checked on a weekly basis by the steering committee. They will receive and evaluate data on inclusion rate and the primary end point event rate. Further, the steering committee will receive and evaluate the weekly safety data on the rate of stent thrombosis in the three groups.

Statistics and data management:

* The statistical analyses will be performed by UNI-C, Aarhus.
* Primary end point. The composite end point in the two groups at six month follow-up will be described by Kaplan-Meier event graphs. The event graphs in the two groups will be compared by a log-rank test. A two-sided test is used. A p-value of < 0.05 is considered significant.
* Secondary end points and other variables. For continuous variables, differences between the treatment groups will be evaluated by Wilcoxon's rank-sum test. For discrete variables, differences will be expressed as counts and in percent and will be analyzed with the chi-square or Fisher's exact test. Secondary end points will be assessed after 6 or 8 months. Two- sided test is used and the p-value considered indicating significance will be 0.05.

Safety:

* For safety reasons, stent thrombosis after one month will be monitored continuously. A stent thrombosis rate of > 5% in any of the treatment groups will necessitate premature termination of the study.

Analysis population:

* The results will be analyzed according to the intention-to-treat principle, i.e. patients randomized to a certain group will be followed and assessed irrespectively of the actual treatment. Protocol violations will be noted and the responsible centres notified.

Sample size calculation:

* A total of 225 patients will be included in each group, in total 450 patients. This is based on the following: We expect a MACE rate of 2% in the group of dilatation of side branch through main vessel stent and of 8% in the group without side branch dilatation through main vessel stent. With an alfa of 5% and a strength of 80%, 206 patients will be needed in each group (two-sided chi square test) to demonstrate this difference. By including 225 patients in each group, a possible dropout before follow-up is counted for.

Randomization procedure:

* The patient will be randomized after successful stenting of the main vessel. There will be a block randomization according to country and a stratification according to sex, age > 70 years, diabetes, +/- measurement of FFR and +/- angiographic follow-up. The patients will be computer randomized by a 24 hour telephone service.

Monitoring of the study:

* The study will be monitored according to the GCP rules by independent professionals.

Publication:

* Results, positive as well as negative, will be published in an international cardiovascular journal. Publication and author issues will be decided by the steering committee on basis of general involvement in the study (core lab. function, end point committee membership etc.) and of number of included patients.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable angina pectoris. -Bifurcation lesion of "LAD/diagonal", "Cx/obtuse marginal", "RCA--
* PDA/posterola¬te¬ral branch" or "LM/Cx/LAD".
* Diameter of main vessel by visual estimate > 2.5 mm.
* Diameter of side branch by visual estimate > 2.25 mm.
* Signed informed consent

Exclusion Criteria:

* Age < 18 years.
* ST-elevation infarction within 24 hours.
* Expected survival < 1 year.
* S-creatinine > 200 µmol/l.
* Allergy to Aspirin, Clopidogrel or Ticlopidine.
* Allergy to Sirolimus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 477 (Actual)
Dates: Start 2007-04-02 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Combined end point of: cardiac death, index lesion myocardial infarction, stent thrombosis or target lesion revascularisation | After 6 months

SECONDARY OUTCOMES:
MACE (cardiac death, myocardial infarction, stent thrombosis or target vessel revascularisation) | during hospital period, after 1, 8, and 14 months, 2 and 3 years
Cardiac death | during hospital period, after 1, 8 and 14 months, 2 and 3 years
Myocardial infarction | during hospital period, after 1, 8 and 14 months, 2 and 3 years
Stent thrombosis | during hospital period, after 1, 8 and 14 months, 2 and 3 years
Target vessel revascularisation | during hospital period, after 1, 8 and 14 months, 2 and 3 years
Total mortality | during hospital period, after 1, 6, 8 and 14 months, 2 and 3 years
Target lesion revascularisation | during hospital period, after 1, 8 and 14 months, 2 and 3 years
Myocardial infarction | related to the index procedure
CCS angina score | after 1, 8 and 14 months, 2 and 3 years
Angiographic significant stenosis (>50%) of main vessel and/or occlusion of the side branch | after 8 months
Late loss of main vessel and side branch | after 8 months
Angiographic significant stenosis (>50%) of main vessel and/or side branch | after 8 months
Angiographic significant stenosis (>50%) of main vessel | after 8 months
Angiographic significant stenosis (>50%) of side branch | after 8 months
Markers | before and after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Niels R Holm, MD, Principal Investigator — MD
Locations (1):
- Aarhus University Hospital Skejby, Aarhus, Denmark

REFERENCES:
- [Derived] Niemela M, Kervinen K, Erglis A, Holm NR, Maeng M, Christiansen EH, Kumsars I, Jegere S, Dombrovskis A, Gunnes P, Stavnes S, Steigen TK, Trovik T, Eskola M, Vikman S, Romppanen H, Makikallio T, Hansen KN, Thayssen P, Aberge L, Jensen LO, Hervold A, Airaksinen J, Pietila M, Frobert O, Kellerth T, Ravkilde J, Aaroe J, Jensen JS, Helqvist S, Sjogren I, James S, Miettinen H, Lassen JF, Thuesen L; Nordic-Baltic PCI Study Group. Randomized comparison of final kissing balloon dilatation versus no final kissing balloon dilatation in patients with coronary bifurcation lesions treated with main vessel stenting: the Nordic-Baltic Bifurcation Study III. Circulation. 2011 Jan 4;123(1):79-86. doi: 10.1161/CIRCULATIONAHA.110.966879. Epub 2010 Dec 20. PMID 21173348
- See also: Publication, primary outcome — http://circ.ahajournals.org/content/123/1/79.long